CLINICAL TRIAL: NCT00543400
Title: A Randomized, Open-label, Parallel Group Feasibility Study to Determine the Safety and Efficacy of M118 vs. Unfractionated Heparin (UFH) in Subjects With Stable Coronary Artery Disease Undergoing Percutaneous Coronary Intervention (PCI)
Brief Title: Evaluation of M118 in Percutaneous Coronary Intervention (EMINENCE)
Acronym: EMINENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOM-M118-006
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Percutaneous Coronary Intervention (PCI)
MeSH Terms: conditions — Coronary Artery Disease | interventions — M-118 compound; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 70 U/kg of unfractionated heparin given IV (Active Comparator): Venous injection (IV) of 70 units per kilogram (U/kg) of unfractionated heparin prior to percutaneous coronary intervention. If procedure lasts longer than 30 minutes a 1/2 rebolus of the original therapy will be given.
  Interventions: Drug: Unfractionated Heparin
- 50 IU/KG of M118 (Experimental): Venous injection of 50 international units per kilogram (IU/kg) of M118 prior to percutaneous coronary intervention. If procedure lasts longer than 30 minutes a 1/2 rebolus of the original therapy will be given.
  Interventions: Drug: M118
- 75 IU/KG of M118 (Experimental): Venous injection of 75 IU/kg of M118 prior to percutaneous coronary intervention. If procedure lasts longer than 30 minutes a 1/2 rebolus of the original therapy will be given.
  Interventions: Drug: M118
- 100 IU/KG of M118 (Experimental): Venous injection of 100 IU/kg of M118 prior to percutaneous coronary intervention. If procedure lasts longer than 30 minutes a 1/2 rebolus of the original therapy will be given.
  Interventions: Drug: M118

INTERVENTIONS:
Drug: M118 — intravenous (IV) infusion
  Arms: 100 IU/KG of M118; 50 IU/KG of M118; 75 IU/KG of M118
Drug: Unfractionated Heparin — IV infusion
  Arms: 70 U/kg of unfractionated heparin given IV

SUMMARY:
The primary objective is to evaluate the safety and feasibility of using M118 as an anticoagulant in the target population of subjects with stable coronary artery disease (CAD) undergoing percutaneous coronary intervention (PCI).

The secondary objectives are to evaluate the effect of M118 on procedural indices including procedure success, abrupt closure, post-procedure TIMI flow, and catheter thrombus.

Substudy Primary Objective The primary objective of the substudy is to characterize the pharmacokinetic and pharmacodynamic profile of M118 among subjects with stable coronary artery disease undergoing elective PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years
* Ability to give informed consent
* Documented stable CAD with a significant lesion in a native coronary artery amenable to PCI with one stent
* Planned single vessel intervention

Exclusion Criteria:

* Myocardial infarction or unstable angina within the prior 7 days
* Target lesion is a chronic total occlusion (present for longer than 3 months)
* Target lesion with angiographically visible thrombus or in-stent thrombosis
* Target lesion is in a bypass graft
* Planned use of a GP IIb/IIIa inhibitor or planned use of atherectomy including directional, rotational, or laser
* Known allergies or sensitivities to heparin, pork, or pork-containing products
* History of HIT
* Hemodynamic instability
* Stroke or Transient Ischemic Attack (TIA) in the prior 3 months
* Active bleeding or bleeding diathesis
* Trauma or major surgery in the preceding month or planned surgery or PCI within the 30 days after the index PCI
* Suspected aortic dissection
* Receiving oral anticoagulation therapy
* Receipt of LMWH or of UFH (except for that used during the diagnostic portion of the index procedure) within the prior 7 days
* ACT > 200 prior to study drug administration
* Severe, untreated hypertension at the time of the index PCI procedure (systolic blood pressure of > 180 mm Hg, diastolic blood pressure > 90 mm Hg)
* Hemoglobin level of less than 10.0 g/dl or a hematocrit below 30%
* Platelet count of less than 100,000 per cubic millimeter or more than 600,000 per cubic millimeter
* Creatinine clearance < 30 mL/min
* Any malignancy within the prior 5 years with the exception of non-melanoma skin cancers
* Prior enrollment in EMINENCE trial or currently receiving other experimental therapy
* Pregnant or lactating if subject is female

Substudy:

Inclusion:

* Ability to give informed consent
* Participation in the main study protocol

Exclusion:

-Inability to provide the blood specimens required by the substudy protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Rao, MD, Principal Investigator — Duke Clinical Research Institute
Locations (44):
- United States (37):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Washington Hospital Center, Medstar Research Institute, Washington D.C., District of Columbia
  - Jim Moran Heart & Vascular Research Institute, Fort Lauderdale, Florida
  - Shands Jacksonville Medical Center (UFL), Jacksonville, Florida
  - Cardiology Research Associates, Ormond Beach, Florida
  - Suncoast Cardiovascular Research, St. Petersburg, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Advocate Good Shephard Hospital, Barrington, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Trinity Medical Center, Rock Island, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Kentucky-Gill Heart Institute, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Hospital Heart & Vascular Institute, Detroit, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Saint Mary's Duluth Clinic Health Center, Duluth, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Saint-Luke's Hospital / Mid America Heart Institute, Kansas City, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - UNC Health Systems, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - Genesis Health Care System, Zanesville, Ohio
  - Allegheny Hospital, Pittsburgh, Pennsylvania
  - Black Hills Clinical Research Center, Rapid City, South Dakota
  - Centennial Heart Cardiovascular Consultants, Nashville, Tennessee
  - Northwest Texas Healthcare System_Amarillo Heart Clinical Research Institute, Inc., Amarillo, Texas
  - Austin Heart, P.A., Austin, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - The Methodist Hospital, Houston, Texas
  - Victoria Heart & Vascular Center, Victoria, Texas
  - Providence Health Center, Waco, Texas
  - UVA Cardiology, UVA Health System, Charlottesville, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Comprehensive Cardiology Care, Milwaukee, Wisconsin
- Canada (7):
  - University of Alberta Hospital, WMC, Edmonton, Alberta
  - Vancouver General Hospital: Interventional Research, Vancouver, British Columbia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec

REFERENCES:
- [Background] Melloni C, Fier I, Roach J, Kosinski AS, Broderick S, Sigmon K, Myles S, Becker RC, Rao SV; EMINENCE Investigators. Design and rationale of the Evaluation of M118 IN pErcutaNeous Coronary intErvention (EMINENCE) trial. Am Heart J. 2009 Nov;158(5):726-33. doi: 10.1016/j.ahj.2009.08.020. Epub 2009 Sep 30. PMID 19853689
- [Result] Rao SV, Melloni C, Myles-Dimauro S, Broderick S, Kosinski AS, Kleiman NS, Dzavik V, Tanguay JF, Chandna H, Gammon R, Rivera E, Alexander JH, Fier I, Roach J, Becker RC; EMINENCE Investigators. Evaluation of a new heparin agent in percutaneous coronary intervention: results of the phase 2 evaluation of M118 IN pErcutaNeous Coronary intErvention (EMINENCE) Trial. Circulation. 2010 Apr 20;121(15):1713-21. doi: 10.1161/CIRCULATIONAHA.109.913277. Epub 2010 Apr 5. PMID 20368520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 503 patients undergoing elective percutaneous coronary intervention at 43 centers in the United States and Canada were randomized
Period: Overall Study
Arm/Group | 70 U/kg of Unfractionated Heparin Given IV | 50 IU/kg of M118 | 75 IU/KG of M118 | 100 IU/kg of M118
Started | 151 | 44 | 152 | 156
Completed | 146 | 43 | 148 | 151
Not Completed | 5 | 1 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 70 U/kg of Unfractionated Heparin Given IV | 50 IU/KG of M118 | 75 IU/KG of M118 | 100 IU/KG of M118 | Total
Number analyzed (Participants) | 151 | 44 | 152 | 156 | 503
Age, Continuous [Mean (Full Range); unit: years] — Overall age of participants
  years | 63.8 [56.8 to 71.6] | 62.9 [54.1 to 70.9] | 65.3 [57.4 to 71.0] | 63.0 [58.3 to 69.9] | 63.9 [54.1 to 71.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 13 | 44 | 47 | 139
  Male | 116 | 31 | 108 | 109 | 364

OUTCOME MEASURES:

1. Primary Outcome: Clinical Events Defined as the Composite of 30-day Death, MI, Repeat Revascularization, Catheter Thrombus, Stroke, Thrombocytopenia, Bailout Use of Glycoprotein IIb/IIIa Inhibitors and Bleeding.
Time Frame: 30 days
Measure: Number; unit: patients experiencing an event
Arm/Group | 70 U/kg of Unfractionated Heparin Given IV | 50 IU/kg of M118 | 75 IU/KG of M118 | 100 IU/kg of M118
Number analyzed (Participants) | 151 | 44 | 152 | 156
patients experiencing an event | 47 | 10 | 43 | 47

ADVERSE EVENTS:
Groups:
- 70 U/kg of Unfractionated Heparin Given IV: Venous injection of 70 units per kilogram (U/kg) of unfractionated heparin prior to percutaneous coronary intervention. If procedure lasts longer than 30 minutes a 1/2 rebolus of the original therapy will be given.
Arm/Group | 70 U/kg of Unfractionated Heparin Given IV | 50 IU/kg of M118 | 75 IU/KG of M118 | 100 IU/kg of M118
Serious Adverse Events (participants affected / at risk) | 20/151 | 5/44 | 15/152 | 15/156
Other Adverse Events (participants affected / at risk) | 116/151 | 36/44 | 116/152 | 114/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 70 U/kg of Unfractionated Heparin Given IV (N=151) | 50 IU/kg of M118 (N=44) | 75 IU/KG of M118 (N=152) | 100 IU/kg of M118 (N=156)
All Serious Adverse Events (General disorders) | 20 | 5 | 15 | 15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 70 U/kg of Unfractionated Heparin Given IV (N=151) | 50 IU/kg of M118 (N=44) | 75 IU/KG of M118 (N=152) | 100 IU/kg of M118 (N=156)
Catheter site hematoma (Injury, poisoning and procedural complications) | 20 | 2 | 22 | 28
Catheter site pain (Injury, poisoning and procedural complications) | 11 | 2 | 12 | 17
Catheter site hemorrhage (Injury, poisoning and procedural complications) | 8 | 2 | 6 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 11 | 17 | 18
Noncardiac chest pain (General disorders) | 10 | 4 | 7 | 14
Nausea (Gastrointestinal disorders) | 13 | 3 | 10 | 16
Angina pectoris (Cardiac disorders) | 14 | 5 | 12 | 10
Headache (Nervous system disorders) | 16 | 1 | 11 | 13
Dizziness (Nervous system disorders) | 6 | 4 | 9 | 7
Hypotension (Vascular disorders) | 9 | 2 | 11 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes